CLINICAL TRIAL: NCT03423368
Title: Assessment of the Effects of Policaptil Gel Retard® on the Glycemic, Lipid and Weight Profile in Overweight and Mild Obese Subjects
Brief Title: Policaptil Gel Retard® in Overweight and Mild Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POLI-14-1
Record Dates: First submitted 2018-01-15; First posted 2018-02-06 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Overweight and Obesity
Keywords: Libramed; Policaptil Gel Retard; Overweight; Obesity; Medical Device; glycemic profile; lipid profile
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Libramed (Experimental): Each patient will be admistered 6 tablets/day (3 tablets before lunch, 3 tablets before dinner) of Libramed for 30 days
  Interventions: Device: Libramed
- Placebo (Placebo Comparator): Each patient will be admistered 6 tablets/day (3 tablets before lunch, 3 tablets before dinner) of placebo for 30 days
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Libramed — Policaptil Gel Retard
  Arms: Libramed
Device: Placebo — Placebo-comparator
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled, interventional clinical study aimed at evaluating the effects of the medical device Libramed (Policaptil Gel Retard®) on the glycemic, lipid and weight profile in overweight and mild obese subjects

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, interventional clinical study on a medical device Visit schedule V1 (day -25) - Screening Visit During this visit (V1) the Investigator will collect information regarding the medical history, the demography, the concomitant medications. The eligibility criteria (inclusion and exclusion criteria) will be verified and during this visit the subjects who will meet the eligibility criteria will be enrolled after the signature of the informed consent form. Each subject will be informed verbally and in writing about the nature and all the requirements of the study.

A brief clinical examination will be performed, including evaluation of vital signs (pulse, systolic and diastolic pressure) and anthropometric parameters (body weight, height, BMI, waist circumference, waist-to-hip and waist-to-height ratio).

Blood and urine samples will be collected for safety routine analysis and for specific analysis to test liver and kidney functionality, glycemic and lipid profile (i.e. glycemic / lipid markers values). An Oral Glucose Tolerance Test (OGTT) will be also performed.

A diary will be given to each subject to record their daily food intake (they will be asked to avoid some food and food supplements/ingredients) and physical activity.

The next visit will be scheduled after 15 days. V2 (day -10) - postprandial metabolic profile short-term assessment - Policaptil Gel Retard® intake During this visit the Investigators will perform a brief clinical examination evaluating pulse, systolic and diastolic pressure and anthropometric parameters; a confirmation of eligibility will take place, on the basis of laboratory tests results.

A blood sample will be collected (t0) and then, after the intake of a standard dosage of Libramed®, a standard meal will be supplied. In order to record the postprandial metabolic profile blood samples will be collected 8 times: 30, 60, 90, 120, 150, 180, 240 and 300 minutes after the meal (t1, 2, 3, 4, 5, 6, 7 and 8) to evaluate the postprandial glycemic and lipid profile.

For the first 10 subjects enrolled additional 2 ml of blood will be collected to evaluate VLDL, IDL, LDL, HDL by Density Gradient Ultracentrifugation (DGU). This analysis will be performed at Clinica Medica I, Azienda Ospedaliera di Padova.

Information on adverse events and concomitant medications will be collected and recorded by the investigators.

The subjective appetite will be assessed using 100mm VASs that will have to be completed before Libramed®, before meal and 150 minutes after consumption of meal.

The next visit will be scheduled after 10 days. V3 (day 0) - postprandial metabolic profile short-term assessment - placebo and baseline / randomization During this visit the Investigators will perform a brief clinical examination evaluating pulse, systolic and diastolic pressure and anthropometric parameters; whole-body fat mass (through DXA technique) will be also evaluated.

A blood sample will be collected (t0) and then, after the intake of a standard dosage of placebo, a standard meal will be supplied. In order to record the postprandial metabolic profile blood samples will be collected 8 times: 30, 60, 90, 120, 150, 180, 240 and 300 minutes after the meal (t1, 2, 3, 4, 5, 6, 7 and 8) to evaluate the postprandial glycemic and lipid profile.

For the first 10 subjects enrolled additional 2 ml of blood will be collected to evaluate VLDL, IDL, LDL, HDL by Density Gradient Ultracentrifugation (DGU).

Moreover a blood sample will be collected in the fasting state for specific analysis to test liver and kidney functionality.

The subjective appetite will be assessed using 100mm VASs that will have to be completed before Libramed® or placebo, before meal and 150 minutes after consumption of meal.

All eligible subjects will be randomized to Policaptil Gel Retard® or placebo and a diet to be followed will be given and explained by a dietitian to all the participants. The daily dietary intake of participants during the intervention period will be set to 1200, 1500 or 1800 Kcal/day depending on the nutritional need of each participant (basal energy expenditure), calculated by means of the Harris Benedict equation (see the protocol for details). They will be asked also to make a daily walk (7000-10000 steps average, to be counted by a pedometer that they will be given too).

The subjects will be given enough study product, according to randomization, to reach the following visit. Moreover a new diary will be given to each subject and the old one will be collected.

Information on adverse events and concomitant medications will be collected and recorded by the investigators.

The next visit will be scheduled after 30 days. V4 (day 30) - end of treatment visit and postprandial metabolic profile long-term assessment - treatment During this visit the Investigators will perform a brief clinical examination evaluating pulse, systolic and diastolic pressure and anthropometric parameters; whole-body fat mass (through DXA technique) will be also evaluated.

A blood sample will be collected (t0) and then, after the intake of a standard dosage of placebo or Policaptil Gel Retard®, according to randomization, a standard meal will be supplied. In order to record the postprandial metabolic profile blood samples will be collected 8 times: 30, 60, 90, 120, 150, 180, 240 and 300 minutes after the meal (t1, 2, 3, 4, 5, 6, 7 and 8) to evaluate the postprandial glycemic and lipid profile. Moreover blood samples will be collected in the fasting state for specific analysis to test liver and kidney functionality, for safety routine analysis (also urine sample) and for specific analysis to test liver and kidney functionality.

The subjective appetite will be assessed using 100mm VASs that will have to be completed before Libramed® or placebo, before meal and 150 minutes after consumption of meal.

Information on adverse events and concomitant medications will be collected and recorded by the investigators.

The diaries and all the unused or empty containers of the study products will have to be brought back to the center, in order to evaluate the subject's adherence to the treatment.

A phone call will be scheduled after 7 days. Follow-up (day 37) A phone contact will take place to assess the safety profile (AE/SAE will be evaluated). Information on concomitant medications and a confirmation about dietary restrictions will be collected and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 - 60 years old (18 and 60 included).
* BMI ≥ 25 Kg/m2 and ≤ 34.9 Kg/m2.
* Stable body weight for the 3 months before enrollment.
* Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects.
* Subjects who agree not to alter their diet in any way for the duration of the trial and to maintain it at steady state (according to the forbidden food ingredients or supplements, that have to be avoided, as outlined in the study protocol), apart from the Treatment Period, during which they agree to follow the assigned diet.
* Subjects who agree not to make any major lifestyle changes (e.g. changing their exercise pattern, except as for what specified in the protocol for the Treatment Period) during the trial.
* Consent to the study and willing to comply with all its procedures.
* Postmenopausal women i.e. women who have not experienced a menstrual bleed for a minimum of 12 months or women who have undergone surgical sterilization (tubal closure or ovaries removal). Otherwise, necessity for women of childbearing potential to follow a reliable contraceptive treatment.Contraceptive treatments deemed as reliable for the study purposes are the following: hormonal contraceptives (pill, patch, vaginal ring), intrauterine devices (IUD), subcutaneous implants; barrier systems as condoms or diaphragm and methods based on the recognition of fertility from an hormonal point of view.

Exclusion Criteria:

* Gastrointestinal disorders (i.e. gastric ulcer, Inflammatory Bowel Disease (IBD) / Irritable Bowel Syndrome (IBS)),
* Uncontrolled hypertension (defined as systolic blood pressure ≥180mmHg and / or diastolic blood pressure ≥100mmHg),
* Diabetes as defined by international criteria.
* Chronic liver disease with increased serum transaminase levels (SGOT and / or SGPT > 2 UNL).
* Thyroid disorders (i.e. hyperthyroidism or hypothyroidism).
* Impaired renal function defined as estimated glomerular filtration rate (e-GFR) <60mL/min/1.73m2 according to Modification of Diet in renal Disease (MDRD) formula due to kidney failure or kidney disease / disorders.
* Blood disorders (i.e. anemia) or subjects who donated their blood within 1 month prior to enrolment or had an important blood loss.
* Any chronic disorder or severe disease which, in the opinion of the investigator, might jeopardise subject's safety, compliance with the protocol and/or ability to complete the study.
* Previous gastrointestinal surgery except for appendectomy, hernia surgery, polypectomy, biopsies, colonic and gastric endoscopy.
* History of alcohol, drug or medication abuse.
* Known hypersensitivity or intolerance to the ingredients contained in the test product or the placebo; celiac subjects.
* Female subjects breastfeeding, pregnant, or planning to become pregnant during the duration of the study.
* History of eating disorder (anorexia, bulimia, binge eating disorder).
* Subjects who have taken anti-obesity medication (Orlistat) or food supplements or natural health products taken with the aim to lose weight over the 2 months prior to entry into the study.
* Prokinetic drugs cannot be started during the study period (included the follow-up period).
* The following treatments cannot be started during the study period (included the follow-up period) and the treatment with one of these treatments should be started at least 3 months prior to the beginning of the study at a stable dosage: - pharmacological treatment for dyslipidemia [(3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (the "statins"), fibrates (gemfibrozil, clofibrate and fenofibrate), niacin/nicotinic acid, bile acid binding resins (colestipol and cholestyramine)], antidepressant such as fluoxetine and bupropion, diuretics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in the postprandial glycemic profile - V4 versus V3 - OGTT | day 30 Vs. day 0
  OGTT
Assessment of changes in the postprandial glycemic profile - V4 versus V3 - fasting insulin | day 30 Vs. day 0
  HOMA index and HbA1c values evaluation
Assessment of changes in the postprandial glycemic profile - V4 versus V3 - HOMA index | day 30 Vs. day 0
  HOMA index
Assessment of changes in the postprandial glycemic profile - V4 versus V3 - HbA1c | day 30 Vs. day 0
  HbA1c

SECONDARY OUTCOMES:
Postprandial lipid profile - V4 versus V3 | day 30 Vs. day 0
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, Apo-B
Postprandial glycemic profile after a single consumption of the product - V2 versus V3 - OGTT | day -10 Vs. day 0
  OGTT
Postprandial glycemic profile after a single consumption of the product - V2 versus V3 - fasting insulin | day -10 Vs. day 0
  fasting insulin
Postprandial glycemic profile after a single consumption of the product - V2 versus V3 - HOMA index | day -10 Vs. day 0
  HOMA index
Postprandial glycemic profile after a single consumption of the product - V2 versus V3 - HbA1c | day -10 Vs. day 0
  HbA1c
Postprandial lipid profile after a single consumption of the product - V2 versus V3 | day -10 Vs. day 0
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, Apo-B
Anthropometric parameters - body weight | day 30 Vs. day 0
  body weight
Anthropometric parameters - BMI | day 30 Vs. day 0
  body mass index - BMI
Anthropometric parameters -Waist circumference | day 30 Vs. day 0
  Waist circumference
Anthropometric parameters - waist-to-hip ratio | day 30 Vs. day 0
  waist-to-hip ratio
Anthropometric parameters - waist-to-height ratio | day 30 Vs. day 0
  waist-to-height ratio
Systolic /diastolic blood pressure - V4 versus V3 | day 30 Vs. day 0
  Assessment of changes in the systolic /diastolic blood pressure - V4 versus V3 - comparison between groups
Dual energy X-ray absorptiometry - V4 versus V3 | day 30 Vs. day 0
  Measurement of whole-body fat mass, through dual energy X-ray absorptiometry (DXA) technique (Noakes et al., 2006; Frestedt et al., 2008) - V4 versus V3 - comparison between groups
Feeling of hunger and feeling of appetite - V4 versus V3 | day 30 Vs. day 0
  100-mm Visual Analog Scale (VAS) evaluation. From 0 (very strong hunger feeling) to 100 (very weak hunger feeling)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.aboca.com/it/i-nostri-prodotti/fitomagra-libramed